CLINICAL TRIAL: NCT05128474
Title: Effectiveness of The Neuromuscular Control-Based Exercise Training in the Treatment of Partial-Thickness Rotator Cuff Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ezgi Turkmen, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulUC49
Record Dates: First submitted 2021-10-22; First posted 2021-11-22 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Rotator Cuff Tear or Rupture, Not Specified as Traumatic; Pain, Shoulder
Keywords: Rotator Cuff Tear; Physiotherapy; Rehabilitation; Neuromuscular Control; Rupture
MeSH Terms: conditions — Rotator Cuff Injuries; Rupture; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Neuromuscular Control-Based Exercise Training Group
  Interventions: Other: Neuromuscular Control-Based Exercise Training Group
- Group 2 (Active Comparator): Conventional Exercise Training Group
  Interventions: Other: Conventional Exercise Training Group

INTERVENTIONS:
Other: Neuromuscular Control-Based Exercise Training Group — Exercises for the neuromuscular control of the shoulder will be progressed by starting with the body weight, and in the following phases, a program that progresses to exercises that will improve the dynamic stabilization, coordination and proprioception of the shoulder will be applied to train the sensorimotor system. The exercise program will be performed twice a week for 8 weeks (16 sessions).
  Arms: Group 1
Other: Conventional Exercise Training Group — In this group, which will mainly benefit from conventional open kinetic chain strength exercises, a strengthening exercise program will be applied by advancing from body weight to elastic bands and weights. The exercise program will be performed twice a week for 8 weeks (16 sessions).
  Arms: Group 2

SUMMARY:
The aim of this study is to determine and compare the effects of neuromuscular control exercises for the shoulder, and standard conservative exercise programs, which are different forms of exercise and have an important role in the treatment of partial thickness rotator cuff tears on treatment. Thus, it is aimed to compare these exercise types with different mechanisms on treatment, to determine the place of neuromuscular control exercises in treatment and whether they are more effective than conventional exercises.

DETAILED DESCRIPTION:
Rotator cuff (RC) tear shows different symptoms or sometimes can progress asymptomatic. The most common symptoms associated with rotator cuff tears are loss of shoulder range of motion (ROM), shoulder pain exacerbated by overhead activities, nocturnal pain, shoulder dysfunction, and functional limitations. Conservative treatment is the first and most preferred procedure in the treatment of partial tears. Conservative treatment includes patient education, activity modifications, medication, and physiotherapy and rehabilitation programs. In the literature search, it is seen that the studies on the conservative treatment of partial RC tears often include open kinetic chain-weighted standard exercises and strengthening exercise types. It is seen that stabilization and proprioception-based neuromuscular control exercises of the shoulder, which have an important role in restoring neuromuscular control, which is reported to be impaired in shoulder pathologies, are included in some studies and these exercises are generally added to standard treatment. However, it is not known whether neuromuscular control exercises are more effective than other exercises in the standard rehabilitation programs as a result of the combined application of these exercises in this patient group. For this purpose, it is aimed to compare the treatment efficacy of a group consisting of neuromuscular control exercises for the shoulder and a group consisting of conventional exercises and to determine the place of neuromuscular control exercises in treatment.

ELIGIBILITY:
Inclusion Criteria:

* Forty years of age or older patients that had been diagnosed for a partial rotator cuff tear that was unrelated to trauma by a specialist orthopedist with MRI and physical examination and no other shoulder problems on the diagnosed shoulder were included into this study.

Exclusion Criteria:

* Patients diagnosed with full-thickness or massive rotator cuff tear, patients who had undergone previous surgery, patients diagnosed with frozen shoulder or glenohumeral instability, and athletic patients younger than 40 years of age with symptoms of acute RC tear were not included in this study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Constant-Murley Score | The Constant Murley Score assessment will be done between two time points: first time at baseline and second time after 8-weeks rehabilitation program. After treatment, "change" will be evaluated.
  The Constant Murley Score is a 100-point scale consisting of 15 points for pain, 20 points for daily activities, 40 points for pain-free range of motion, and 25 points for strength. High scores are positively correlated with the increased functional level. While pain and activities of daily living are evaluated by the patient, range of motion and strength are evaluated by the clinician.

SECONDARY OUTCOMES:
The Numerical Pain Rating Scale (NPRS) | Evaluations will be done between two time points: first time at baseline and second time after 8-weeks rehabilitation program. After treatment, "change" will be evaluated.
  The levels of pain felt at rest / activity / night were measured using Numerical Pain Rating Scale (NPRS). Patients were asked to evaluate their pain status with a 10-point scale and high scores are positively correlated with pain.
Shoulder Joint Proprioception with Inclinometer | Evaluations will be done between two time points: first time at baseline and second time after 8-weeks rehabilitation program. After treatment, "change" will be evaluated.
  Proprioception of the shoulder joint is assessed by reproduction/reposition testing using an inclinometer. The patient will be evaluated by recording the difference between the angle from which the patient comes and the target angle determined.
Shoulder Joint Range of Motion (ROM) | Evaluations will be done between two time points: first time at baseline and second time after 8-weeks rehabilitation program. After treatment, "change" will be evaluated.
  The shoulder flexion, abduction, internal and external rotation ROM were evaluated with goniometer while the patient was in supine position.
Shoulder Joint Muscle Strength | Evaluations will be done between two time points: first time at baseline and second time after 8-weeks rehabilitation program. After treatment, "change" will be evaluated.
  Maximum isometric shoulder flexion, abduction, external and internal rotation strength measurements will be performed using a handheld dynamometer. During the test, while the participants were in a sitting position to measure shoulder flexion and abduction forces; for the measurement of external and internal rotational forces in the supine position, the shoulder is in 90° abduction and the elbow is in 90° flexion. For each movement, the measurements are repeated 3 times and the best measurement value is recorded.
Quick DASH (Disabilities of the Arm, Shoulder and Hand) Questionnaire | Evaluations will be done between two time points: first time at baseline and second time after 8-weeks rehabilitation program. After treatment, "change" will be evaluated.
  Quick DASH is a 11-item questionnaire that questions the activities of a person in daily life, the degree of participation in recreational activities, the symptom and psychosocial state that affects their pain, and sleep quality. The total score is at least 0 and at most 100, and the high scores are positively correlated with the decreased functional level.
Short Form 12 (SF-12) | Evaluations will be done between two time points: first time at baseline and second time after 8-weeks rehabilitation program. After treatment, "change" will be evaluated.
  SF-12 was used to assess physical and mental health-related quality of life. The total score is at least 0 and at most 100, and the high scores are positively correlated with high quality of life.
Global Rating of Change (GRC) Scale | Evaluations will be done between two time points: first time at baseline and second time after 8-weeks rehabilitation program. After treatment, "change" will be evaluated.
  Global Rating of Change (GRC) scale was used to assess the overall satisfaction levels of the patients. Patients were asked to evaluate their post-treatment status with a 5-point likert scale and high scores are positively correlated with satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Üniversitesi-Cerrahpaşa, Sağlık Bilimleri Fakültesi, Istanbul, Büyükçekmece, Turkey (Türkiye)